CLINICAL TRIAL: NCT01702584
Title: Efficacy and Safety of StENt-assisted Treatment for CErebral Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kobe City General Hospital (Other)
Responsible Party: Principal Investigator, Nobuyuki Sakai, Director of Neurosurgery, Kobe City General Hospital
Other Study IDs: TRIBRAIN1204; UMIN000010405 (Other: UMIN Japan)
Record Dates: First submitted 2012-09-05; First posted 2012-10-08 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stent Embolisation
Keywords: stent; intracranial aneurysm; embolization; adverse event
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stent assisted embolization: stent assisted embolization of intracranial aneurysm
  Interventions: Procedure: stent assisted embolization

INTERVENTIONS:
Procedure: stent assisted embolization — stent assisted embolization and anti-thrombotic management
  Other Names: Enterprise VRD

SUMMARY:
Prospective registry study to evaluate safety and efficacy of stent assisted embolization of intracranial aneurysm.

DETAILED DESCRIPTION:
To evaluate stent assisted embolization of intracranial aneurysm, record information about treatment and any event (death, stroke, hemorrhagic event) prospectively.

ELIGIBILITY:
Inclusion Criteria:

* stent assisted embolization of intracranial aneurysm
* 20 or more year old

Exclusion Criteria:

* not determined

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stent assisted embolization of intracranial aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
any death, stroke and major hemorrhagic event | 2 years after treatment
  any death, stroke and major hemorrhagic event within 2 years after treatment

SECONDARY OUTCOMES:
any adverse event | 2 years
  1. death, stroke, hemorrhagic event within 30days or between 31days to 2years after treatment
  2. any change of anti-thrombotic therapy within 2years after treatment
  3. recanalization or re-treatment within 2years after treatment
  4. stent stenosis or occlusion within 2years after treatment
  5. any adverse event within 2years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sakai, MD, DMSc, Principal Investigator — Kobe City Medical Center General Hospital
Locations (1):
- Kobe City Medical Center General Hospital, Kobe, Hyōgo, Japan